CLINICAL TRIAL: NCT01269827
Title: Randomized, Double-Blinded, Controlled Clinical Trial of the Effect Pentoxifylline vs Placebo on the Serum Concentrations of TNF-a, IL-6 and CRP of Patients in Hemodialysis
Brief Title: Pentoxifylline and Systemic Inflammation in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Alfonso Martín Cueto Manzano, Jefe de Unidad de Investigación Médica en Enfermedades Renales, HE, CMNO, IMSS, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-1A-I-007; other grant (Other Grant/Funding Number: Fondo de Fomento a la Investigación (No. 2006-1A-I-007))
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Inflammation; End-stage Renal Disease; Hemodialysis
Keywords: inflammation; pentoxifylline; hemodialysis
MeSH Terms: conditions — Inflammation; Kidney Failure, Chronic | interventions — Pentoxifylline; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pentoxifylline (Experimental)
  Interventions: Drug: Pentoxifylline
- placebo (Placebo Comparator)
  Interventions: Drug: starch tablets

INTERVENTIONS:
Drug: Pentoxifylline — Over a period of 4 months, patients of the study group received one PTX tablet (400 mg) orally once a day (at dinner time)
  Other Names: trental
  Arms: pentoxifylline
Drug: starch tablets — Over a period of 4 months, patients of the control group received one starch tablet orally once a day (at dinner time)
  Other Names: placebo
  Arms: placebo

SUMMARY:
The aim of this study was to compare the effect of PTX vs placebo on serum concentrations of TNF-α, IL-6, and CRP in patients on hemodialysis.

DETAILED DESCRIPTION:
Patients were randomly selected from the total HD patients of our hospital. Once included, patients were randomly allocated (by a computer-generated randomization list) to a study or control group. Over a period of 4 months, patients of the study group received one PTX tablet (400 mg) orally once a day (at dinner time), whereas controls received one starch identical tablet on the same schedule.

All patients had three HD sessions per week, with the same kind of single-use dialysis membrane and dialysate. Monthly visits were scheduled for clinical and biochemical evaluations. A blood sample was taken at baseline and every month for measurement of complete blood count, urea, creatinine, glucose, albumin, lipids, and electrolytes (measured by usual methods). In serum samples at 0, 2 and 4 months, TNF-α and IL-6 concentrations were measured by ELISA using high sensitivity kits (Amersham Pharmacia Biotech, Buckinghamshire, UK). Additionally, in the same serum samples, CRP concentrations were measured by nephelometry using high sensitivity kits (Dade Behring, Marburg, Germany) in a Nephelometry Analyzer II (Dade Behring, Marburg, Germany). All laboratory measurements, including inflammation markers, were performed in the Central Laboratory (Hospital de Especialidades, CMNO), by the same personnel blinded to patient's details.

Treatment compliance was recorded by counting tablets left in the container at the end of each monthly visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years,
* ≥2 months on HD,
* arteriovenous fistula as vascular access, and
* endorsement of informed consent.

Exclusion Criteria:

* inflammatory cause of ESRD,
* liver disease, cancer, AIDS,
* any infectious disease 2 months before the study,
* failed kidney graft,
* hypersensitivity to PTX or other methylxanthines,
* hemorrhage/clotting disorders,
* risk for worsening pre-existing cardiac arrhythmias or arterial hypotension,
* treatment with antibiotics, non-steroidal anti-inflammatory drugs, steroids, immunosuppressives, statins or PTX 3 months previous to the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
serum levels of TNF-a, IL-6 and CRP | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso M. M Cueto-Manzano, MD, MSc, PhD, Study Chair — Unidad de Investigación Médica en Enfermedades Renales, Hospital de Especialidades, CMNO, IMSS
Locations (1):
- Hospital de Especialidades, CMNO, IMSS, Guadalajara, Jalisco, Mexico